CLINICAL TRIAL: NCT05099185
Title: Measurement of Water-soluble Vitamins and Trace Elements Loss With Maintenance Post-dilution Haemodiafiltration Patient
Brief Title: Water Soluble Vitamins and Trace Elements Loss in Hemodiafiltration Patients
Acronym: VITAFLUX
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0491; 2021-A01241-40 (Other: ID-RCB)
Record Dates: First submitted 2021-07-16; First posted 2021-10-29 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Chronic Hemolysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — This study collect and analyse dialysate sample through a device called sampler was developed by the THERADIAL® company. Sampler collect continuously during the dialysis session, one hundred of the effluent liquid (ie a calibrated sample of dialysate) before it is eliminated in the sewer. The dialysate samples will be analyzed by the Lyon Sud biochemistry laboratory immediately after the end of the session
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Maintenance online post-dilution hemodiafiltration patients: Maintenance hemodialysis patients who undergo hemodialysis 3 times per week with online post-dilution hemodiafiltration process
  Interventions: Biological: Water-soluble vitamins and trace elements measures

INTERVENTIONS:
Biological: Water-soluble vitamins and trace elements measures — We would like to measure water-soluble vitamins (B1, B6, B9, B12, C) and trace elements (zinc, selenium) in blood and dialysate for the patients treated by online post-dilution hemodiafiltration patients. There measures on blood are done systematically during the half-yearly report of our patients in our hemodialysis center. Only results are collect for the study.

SUMMARY:
End stage renal disease is a severe pathology in which some toxic waste and an excessive amount of water can accumulate in the human body with life threatening consequences. Maintenance hemodialysis is one of the possible treatment for this disease.

Hemodialysis filter the blood through a membrane according to a dialysis bath and so can be able to purify the blood of the toxic waste.

Otherwise, since the 1980s, the investigator know that patient in maintenance hemodialysis can have some deficiency in water soluble vitamins and trace elements. Mechanisms of the deficiency are multiple (a decreased of food intake, a diminution of the appetite, digestive malabsorption du to medics and comorbidities and loss in hemodialysis).

Impact of this deficiency have an important impact on vital prognosis for these patients. These nutrients are essential for AND synthesis, mechanism of inflammation, cells membranes synthesis, etc. DOPPs study in 2004 have shown a decreased of 16% in the mortality within 4 years with supplemented patients. Also, since this study, international recommendations were wrote in 2009, then in 2020, in order to supplement in vitamins and trace elements patients in maintenance conventional hemodialysis.

Despite these recommendations, some supplementary efforts are necessary, especially since online hemodiafiltration, a new process, is widely available and used in particular in Europe. This process combines 2 phenomena, diffusion and convection, through high-flux membranes. This process can remove a large quantity of molecule present in blood and especially the middle-molecule. In return, a more important quantity of water soluble vitamins and oligo-elements could be removed by this technique.

Also, the investigator would like to measure this loss of vitamins and trace-elements in patients with maintenance online post-dilution hemodiafiltration process with dialysate sample and blood concentrations measured (usual patient monitoring) during the session.

ELIGIBILITY:
Inclusion Criteria:

* Maintenance hemodialysis more than 3 months
* 3 sessions per week during 4 hours
* Hemodiafiltration process used with this patient on Lyon Sud Hospital
* Flow of the vascular access > 300 mL/min at least
* Age > 18 years
* Patient able to understand the study's goal

Exclusion Criteria:

* Active infectious or inflammatory disease
* Active malignant disease
* Intestinal malabsorptive disease
* Polysulfone's dialysis membrane allergy
* Patient under guardianship and judicial protection
* Pregnant and breastfeeding woman
* Opposition to the study

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Maintenance hemodialysis patients who are treated in nephrology unit at Centre Hospitalier de Lyon Sud with online hemodiafiltration process
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Comparison of the blood concentrations measured in vitamins and trace elements before and after the hemodialysis session by the post-dilution HDF technique during the half-yearly assessment (usual patient follow-up). | Day 1
  We would like to measure the concentrations of water-soluble vitamins and trace elements in dialysate by collecting 1% of this by Theraflux® device, and compare to the blood concentration collecting during the half-yearly report at the beginning then at the end of one hemodialysis session with online post-dilution hemodiafiltration session.

CONTACTS AND LOCATIONS:
Overall Officials: Etienne NOVEL-CATIN, MD, Principal Investigator — Nephrology department
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France